CLINICAL TRIAL: NCT02625116
Title: ELENA Cohort: A Long-term Longitudinal Study in a Pediatric Sample With Autism Spectrum Disorders
Acronym: ELENA
Status: Active, not recruiting | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Caisse Nationale de Solidarité pour l'Autonomie (Other)
Responsible Party: Sponsor
Other Study IDs: 8852-2
Record Dates: First submitted 2015-12-04; First posted 2015-12-09 (Estimated); Last update posted 2024-05-28 (Actual); Status verified 2024-05

CONDITIONS: Autism Spectrum Disorders
Keywords: Cohort
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The objective of the ELENA French Cohort is to study the developmental trajectories of children and adolescents with ASD and their risk or protective associated factors.

This is an open, prospective and multicenter cohort study, including children and adolescents under 16 years of age with ASD recruited from services specialized in the assessment of developmental disorders.

DETAILED DESCRIPTION:
Multidisciplinary cohort studies of children with Autism Spectrum Disorders (ASD) followed from childhood to adulthood exist abroad but not in France. The objective of the ELENA French Cohort is to study the developmental trajectories of children and adolescents with ASD and their risk or protective associated factors.

This is an open, prospective and multicenter cohort study, including children and adolescents under 16 years of age with ASD recruited from services specialized in the assessment of developmental disorders. The patients will be monitored every 18 months for at least 36 months and during a maximum of 10 years. Clinical, social, environmental, and genetic data, as well as data relating to the parental quality of life will be collected. The primary endpoint will be the adaptive level in three domains of the Vineland II (Communication, Socialization and Daily living skills). The secondary endpoints will be parental quality of life, comorbidities, interventions and severity of ASD.

The inclusion of 900 patients over a 10-year period is expected. This cohort should contribute to a better knowledge of the child with ASD's development, taking into account his physical, social and familial environment, the type of interventions and some genetic components. It should also lay the foundations for a national network of professionals working in the field of autism research by offering them a common tool for promoting translational studies.

ELIGIBILITY:
Inclusion Criteria:

* Age between 2 and 16 years
* Diagnosis of ASD formally established during a multidisciplinary assessment, according ICD 10 criteria and ADI
* Patient who benefited in the last 12 months: Vineland, ADOS, intellectual level
* Parents consent

Exclusion Criteria:

* Subject refusal to participate
* Parental refusal to participate

Ages: 2 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The study population is aged between 2 and 16 years, and has a diagnosis of ASD formally established during a multidisciplinary assessment and made according international criteria of the ICD10.
Sampling Method: Non-Probability Sample
Enrollment: 919 (Actual)
Dates: Start 2014-09-27 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Adaptive behavior scores obtained using the three sub-scales of the Vineland Adaptive Behavior Scale | 18 months
  Communication, Daily Living Skills and Socialization

CONTACTS AND LOCATIONS:
Overall Officials: Amaria BAGHDADLI, Profesor, Principal Investigator — Autism Ressource Center
Locations (1):
- CHU Montpellier-Hôpital La Colombière, Montpellier, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Peyre H, Baghdadli A. Investigating the ADOS-2 calibrated severity score: insights from the ELENA cohort. Front Child Adolesc Psychiatry. 2026 Jan 12;4:1674226. doi: 10.3389/frcha.2025.1674226. eCollection 2025. PMID 41601706
- [Derived] Rattaz C, Peries M, Pickles A, Baghdadli A. The Impact of Inclusive Education Practices on Students With ASD'S Outcomes: Report From the ELENA French Cohort Study. Autism Res. 2026 Jan 8. doi: 10.1002/aur.70164. Online ahead of print. PMID 41508375
- [Derived] Nemorin H, Michelon C, Peyre H, Monnier M, Peries M, Baghdadli A. Profiling clinical heterogeneity in Autism Spectrum Disorder at time of children's diagnosis: A cluster analysis from the ELENA cohort. Res Dev Disabil. 2025 Aug;163:105040. doi: 10.1016/j.ridd.2025.105040. Epub 2025 May 22. PMID 40409244
- [Derived] Mortamais M, Ongono JS, Michelon C, Hough I, Seyve E, Kloog I, Zaros C, Charles MA, Lepeule J, Baghdadli A. Prenatal Exposure to Ambient Particulate Matter and Autism Spectrum Disorder in Children, a Case Control Study in France. J Autism Dev Disord. 2025 Mar 22. doi: 10.1007/s10803-025-06795-y. Online ahead of print. PMID 40120015
- [Derived] Peries M, Duhr F, Picot MC, Heude B, Bernard JY, Baghdadli A. Breastfeeding is not a risk factor for clinical severity in Autism spectrum disorder in children from the ELENA cohort. Sci Rep. 2023 Jan 16;13(1):816. doi: 10.1038/s41598-022-27040-x. PMID 36646708
- [Derived] Berard M, Peries M, Loubersac J, Picot MC, Bernard JY, Munir K, Baghdadli A. Screen time and associated risks in children and adolescents with autism spectrum disorders during a discrete COVID-19 lockdown period. Front Psychiatry. 2022 Dec 1;13:1026191. doi: 10.3389/fpsyt.2022.1026191. eCollection 2022. PMID 36532191
- [Derived] Dellapiazza F, Michelon C, Rattaz C, Picot MC, Baghdadli A. Sex-related differences in clinical characteristics of children with ASD without ID: Results from the ELENA cohort. Front Psychiatry. 2022 Nov 28;13:998195. doi: 10.3389/fpsyt.2022.998195. eCollection 2022. PMID 36518364
- [Derived] Vernhet C, Michelon C, Dellapiazza F, Rattaz C, Geoffray MM, Roeyers H, Picot MC, Baghdadli A; ELENA study group. Perceptions of parents of the impact of autism spectrum disorder on their quality of life and correlates: comparison between mothers and fathers. Qual Life Res. 2022 May;31(5):1499-1508. doi: 10.1007/s11136-021-03045-3. Epub 2021 Nov 25. PMID 34822048
- [Derived] Miniarikova E, Vernhet C, Peries M, Loubersac J, Picot MC, Munir K, Baghdadli A. Anxiety and depression in parents of children with autism spectrum disorder during the first COVID-19 lockdown: Report from the ELENA cohort. J Psychiatr Res. 2022 May;149:344-351. doi: 10.1016/j.jpsychires.2021.11.022. Epub 2021 Nov 8. PMID 34776249
- [Derived] Berard M, Rattaz C, Peries M, Loubersac J, Munir K, Baghdadli A. Impact of containment and mitigation measures on children and youth with ASD during the COVID-19 pandemic: Report from the ELENA cohort. J Psychiatr Res. 2021 May;137:73-80. doi: 10.1016/j.jpsychires.2021.02.041. Epub 2021 Feb 22. PMID 33662654
- [Derived] Baghdadli A, Miot S, Rattaz C, Akbaraly T, Geoffray MM, Michelon C, Loubersac J, Traver S, Mortamais M, Sonie S, Pottelette J, Robel L, Speranza M, Vesperini S, Maffre T, Falissard B, Picot MC; ELENA Study Group. Investigating the natural history and prognostic factors of ASD in children: the multicEntric Longitudinal study of childrEN with ASD - the ELENA study protocol. BMJ Open. 2019 Jun 19;9(6):e026286. doi: 10.1136/bmjopen-2018-026286. PMID 31221874